CLINICAL TRIAL: NCT05606250
Title: Effectiveness of the Ultrasound-guided Percutaneous Neuromodulation Technique in Post-surgical Anterior Cruciate Ligament Patients
Brief Title: Ultrasound-guided Percutaneous Neuromodulation in Anterior Cruciate Reconstruction
Acronym: NMPeLCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: h8yucsdh
Record Dates: First submitted 2022-10-17; First posted 2022-11-04 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-11

CONDITIONS: ACL Injury
Keywords: percutaneous neuromodulation; femoral nerve; ultrasound; acl reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Control group: The subjects will receive physiotherapy treatment and the experimental group will receive combined treatment of physiotherapy and ultrasound-guided percutaneous neuromodulation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy protocol (No Intervention): The physiotherapy protocol is based on manual therapy (passive joint mobilization), myofascial work, active exercise, high intensity neuromuscular electrical stimulation and cryotherapy.
- Ultrasound-Guided Percutaneous Neuromodulation (Experimental): Ultrasound-guided percutaneous neuromodulation (e-NMP) is the electrical stimulation by means of a needle with ultrasound guidance of a peripheral nerve at some point in its course or of a muscle at a motor point, with a therapeutic purpose.
  The application of the stimulation is carried out with a puncture needle accompanied by a low or medium frequency electrical current.
  In e-MPN, a sensory and/or motor response is sought when the peripheral nerve is stimulated, and a motor response is achieved by stimulating the motor point (uncontrolled exaggerated response that normalizes after the application of the technique).
  Interventions: Other: Ultrasound-Guided Percutaneous Neuromodulation

INTERVENTIONS:
Other: Ultrasound-Guided Percutaneous Neuromodulation — Ultrasound guided percutaneous neuromodulation in femoral nerve. Patients were placed in supine lying with the anterior aspect of the hip uncovered. The intervention consisted of the application of a biphasic square wave electric current, with a frequency of 2 Hz, a phase duration of 250μs, and a maximum tolerable intensity to cause an exacerbated muscle contraction for 15minutes in total
  Arms: Ultrasound-Guided Percutaneous Neuromodulation

SUMMARY:
The objective of the study is to demonstrate the efficacy of the ultrasound-guided percutaneous neuromodulation technique in the femoral nerve in patients who underwent surgery for the anterior cruciate ligament.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all subjects who accept the study and give their informed consent in writing, the subjects will participate in a randomized, longitudinal and prospective clinical trial divided into two groups (control group and experimental group) with the main objective of demonstrating that the ultrasound-guided percutaneous neuromodulation technique is effective for the treatment of pain in subjects undergoing surgery for the anterior cruciate ligament.

Subjects belonging to the control group will perform a physiotherapy protocol and those belonging to the experimental group will undergo two interventions of the ultrasound-guided percutaneous neuromodulation technique combined with the physiotherapy protocol. The same number of measurements will be performed on all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 55 years who have undergone surgery for an anterior cruciate ligament (ACL) in a period of time between 2 and 6 weeks of evolution with or without meniscal injury (meniscal regularization / meniscal suture / meniscectomy, etc.).
* have pain or loss of sensitivity in the operated knee and that they have signed the informed consent.

Exclusion Criteria:

* Subjects with chronic joint disease; prosthesis or osteosynthesis in the intervention area, as well as heart disease, neoplasia and coagulopathy.
* Subjects consuming analgesics.
* Subjects with belonephobia or insurmountable fear of needles
* History of lumbar pathology (lumbar hernia/protrusion) due to possible involvement of the lumbar plexus.
* Subjects with a history of neurological or orthopedic disorders
* Subjects with bilateral symptoms.
* Subjects with epilepsy, pacemaker or pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in pain through the visual analogue scale in 12 weeks | Before treatment, immediately after treatment. Before treatment at week 1 after the first measurement, immediately after treatment at week 1 after the first measurement. Week 4 from the first measurement. Week 12 from the first measurement,
  It allows pain intensity to be measured with maximum reproducibility between observers. It consists of a horizontal line of 10 centimeters, at whose ends are the extreme expressions of a symptom. Absence or less intensity is located on the left and greater intensity on the right. The patient is asked to mark the point on the line that indicates the intensity and it is measured with a millimeter ruler.
  This variable will be measured with a numerical value from 1 to 10.

SECONDARY OUTCOMES:
Changes in DN4 scale en 12 weeks | Before treatment / intervention and week 12.
  The DN4 questionnaire consists of a total of 10 items grouped into 4 sections. The first seven elements are related to the quality of pain (burning, painful cold, electric shocks) and its association with abnormal sensations (pins and needles, tingling, numbness, itching). The other 3 items are related to the neurological examination in the painful area (tactile hypoesthesia, pinprick hypoesthesia, tactile allodynia). A score of 1 is given to each positive element and a score of 0 to each negative element. The total score is calculated as the sum of the 10 items and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.
  This variable will be measured with a numerical value from 1 to 10.
Changes in LEFS scale in 12 weeks | Before treatment / intervention and week 12.
  measure the patient's baseline function, ongoing progress, and functional outcomes. This scale consists of 20 items, and the final score must be between 0 and 80. Items are rated on a 5-point scale, from 0 (extreme difficulty/ inability to perform the activity) to 4 (no difficulty).
  This variable will be measured with a numerical value from 1 to 80.
Changes in range of movement in 12 weeks. | Before treatment, immediately after treatment. Before treatment at week 1 after the first measurement, immediately after treatment at week 1 after the first measurement. Week 4 from the first measurement. Week 12 from the first measurement,
  With goniometry, the patient's flexion and extension will be measured. This variable will be reflected with a numerical value and angle degrees.
Changes in pressure pain threshold in 12 weeks | Before treatment, immediately after treatment. Before treatment at week 1 after the first measurement, immediately after treatment at week 1 after the first measurement. Week 4 from the first measurement. Week 12 from the first measurement,
  Pressure pain threshold (PPT) was assessed with an analog algometer. One point on the epicondyle and five points on both knees (vastus lateralis, vastus medialis, patellar tendon, quadriceps tendon, and hamstring) were evaluated.
  PPT points: (1) 10 cm lateral to the midpoint of the superior border of the patella; (2) 3 cm medial to the midpoint of the superior border of the patella; (3) midway between the inferior border of the patella and the tibial tuberosity; (4) 3 cm proximal to the superior border of the patella; and (5) 3 cm medial to the tibial tuberosity, at the insertion of pes anserinus.
  When the individual reported a change in the sensation of pressure, the value indicated on the algometer was recorded. The subject did not receive information about the values obtained.
  This variable will be reflected with numerical values. The PPT is expressed in kg/m^2 and was measured with an analog algometer.
Changes in heart rate variability in 12 weeks | Before treatment, immediately after treatment. Before treatment at week 1 after the first measurement, immediately after treatment at week 1 after the first measurement. Week 4 from the first measurement. Week 12 from the first measurement,
  The intervals between successive heartbeats (RR intervals) 2 (HRV) domains to detect changes in HRV Time domain (non-spectral): average RR intervals (ms); RMSSD (ms): the square root of the mean value of the sum of the squared differences of all successive R-R intervals; LRMSSD (ms): logarithm of the square root of the mean value of the sum of the squared differences of all successive R-R intervals: SDNN (ms): the standard deviation of the interval between beats from which artifacts were removed (NN); and PNN50: the percentage of differences between adjacent normal R-R intervals of more than 50 ms.
  Frequency domain / spectral measurements (spectral) (HF) and (LF) (ms). minimum, maximum and average heart rate. The subject will be seated for a period of two minutes and thirty seconds. The data will be collected with the BERRY KING HEARTBEAT 2 heart rate meter, and the data will be record.This variable will be reflected with numerical values.
Changes in dynamometry in 12 weeks. | Before treatment, immediately after treatment. Before treatment at week 1 after the first measurement, immediately after treatment at week 1 after the first measurement. Week 4 from the first measurement. Week 12 from the first measurement,
  Dynamometry will be used to assess strength. This variable will be measured with a digital hand dynamometer called the Activ force 2 Digital Dynamometer. The patient will be seated on the stretcher and will actively do three isometric extensions with a 90º angle of knee flexion. This test will be carried out and the maximum extension force data will also be collected between the three knee extensions.
  This variable will be reflected with numerical values.
Body Mass Index | Before treatment / intervention
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Romero Morales, PT, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Julio José Caballero López, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPDs collected
  all IPDs underlying the results of a post
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting in November 2023
Access Criteria: The data obtained through this study can be provided to qualified researchers with an academic interest in percutaneous ultrasound-guided neuromodulation.
URL: https://pubmed.ncbi.nlm.nih.gov

REFERENCES:
- [Background] De-la-Cruz-Torres B, Abuin-Porras V, Navarro-Flores E, Calvo-Lobo C, Romero-Morales C. Ultrasound-Guided Percutaneous Neuromodulation in Patients with Chronic Lateral Epicondylalgia: A Pilot Randomized Clinical Trial. Int J Environ Res Public Health. 2021 May 3;18(9):4877. doi: 10.3390/ijerph18094877. PMID 34063673
- [Background] De-la-Cruz-Torres B, Carrasco-Iglesias C, Minaya-Munoz F, Romero-Morales C. Crossover effects of ultrasound-guided percutaneous neuromodulation on contralateral hamstring flexibility. Acupunct Med. 2021 Oct;39(5):512-521. doi: 10.1177/0964528420920283. Epub 2020 May 13. PMID 32403999
- [Background] Ilfeld BM, Said ET, Finneran JJ 4th, Sztain JF, Abramson WB, Gabriel RA, Khatibi B, Swisher MW, Jaeger P, Covey DC, Robertson CM. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Femoral Nerve for Postoperative Analgesia Following Ambulatory Anterior Cruciate Ligament Reconstruction: A Proof of Concept Study. Neuromodulation. 2019 Jul;22(5):621-629. doi: 10.1111/ner.12851. Epub 2018 Aug 30. PMID 30160335
- [Background] San-Emeterio-Iglesias R, Minaya-Munoz F, Romero-Morales C, De-la-Cruz-Torres B. Correct Sciatic Nerve Management to Apply Ultrasound-Guided Percutaneous Neuromodulation in Patients With Chronic Low Back Pain: A Pilot Study. Neuromodulation. 2021 Aug;24(6):1067-1074. doi: 10.1111/ner.13396. Epub 2021 Apr 20. PMID 33876885
- [Background] Ilfeld BM, Gilmore CA, Grant SA, Bolognesi MP, Del Gaizo DJ, Wongsarnpigoon A, Boggs JW. Ultrasound-guided percutaneous peripheral nerve stimulation for analgesia following total knee arthroplasty: a prospective feasibility study. J Orthop Surg Res. 2017 Jan 13;12(1):4. doi: 10.1186/s13018-016-0506-7. PMID 28086940
- [Derived] Caballero-Lopez J, Navarro-Santana M, Almazan-Polo J, Garcia-Sanz F, Diaz-Arribas MJ, Minaya-Munoz F, Romero-Morales C. Short-term effects of percutaneous electrical nerve stimulation on pain and muscle function in patients undergoing anterior cruciate ligament surgery: a randomized clinical trial. Front Rehabil Sci. 2025 Apr 29;6:1501703. doi: 10.3389/fresc.2025.1501703. eCollection 2025. PMID 40365171